CLINICAL TRIAL: NCT04187092
Title: Knee Biofeedback Rehabilitation Interface for Game-based Home Therapy ("KneeBRIGHT") Phase II
Brief Title: Knee Biofeedback Rehabilitation Interface for Game-based Home Therapy for Patients With Knee Osteoarthritis
Acronym: KneeBRIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Barron Associates, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Hart, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-HSR# 21926
Record Dates: First submitted 2019-11-21; First posted 2019-12-05 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Osteo Arthritis Knee
Keywords: knee osteoarthritis; video-game based interventions; strength; Precision
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants with knee osteoarthritis will be randomly assigned to Group 1 or 2. During each exercise session all the participants will perform stretching exercises, strengthening exercises and balance exercises. Dosage of exercises will be based on the rehabilitation principles and will be guided and progressed the way the participants feel about their knee health throughout the rehabilitation program.
  Participants in Group1 (KneeBright group), will perform some of the exercises with the KneeBright Device and while playing a video game, while Group 2 will undergo standard knee rehabilitation exercises without the KneeBright device.
  Both groups will undergo a 12 week program including 3 exercise sessions per week that include a combination of in-person and at home sessions. Participants in both groups will undergo 36 exercise sessions in total, each lasting for 1 hour. Among these 36 sessions 20 will be performed in clinic under supervision and 16 will be performed at home.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded and will be responsible for executing the baseline and follow-up outcome measures. Assessors have the adequate training and experience for recording the patient reported outcome measures along with conducting the thigh muscle strength and balance testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KneeBright group (Experimental): Participants in this group will perform exercises aimed to improve the muscle strength, balance and precision. Participants will perform exercises three times a week for 12 weeks. Each session will last for an hour. Some of the exercises will be performed with the KneeBright Device while playing a video game.
  Interventions: Other: KneeBright Group
- Standard Rehabilitation group (Active Comparator): Participants in this group will perform exercises with the same focus and frequency. No exercises will be performed with the KneeBright device.
  Interventions: Other: Standard Rehabilitation group

INTERVENTIONS:
Other: KneeBright Group — The KneeBRIGHT group will use KneeBright device which consists of an EMG biofeedback interface software that guides users through exercise routines. The wireless EMG sensors includes two small electrodes that will be made to stick to the quadriceps muscles both sides. KneeBRIGHT software features a virtual world wherein patients complete challenges controlling the in-game avatar with the EMG units during exercises specific to knee osteoarthritis rehabilitation.
  The KneeBRIGHT software will incorporates a variety of exercises for strengthening the quadriceps and will employ algorithms based on the Daily Adjustable Progressive Resistance Exercise (DAPRE) technique, in which the quantity of repetitions performed in these sets is then used to determine the appropriate increase (or possibly decrease) in target resistance for the next sets/sessions.
  Arms: KneeBright group
Other: Standard Rehabilitation group — Participants in this group will undergo standard clinic based knee rehabilitation. Both groups will perform exact same exercises, however, no KneeBRIGHT device will be used in this group.
  Arms: Standard Rehabilitation group

SUMMARY:
Osteoarthritis (OA) is the leading cause of disability in the United States. As osteoarthritis is associated with the lower limb muscle weakness, rehabilitation through quadriceps strengthening is a well-established treatment for patients with knee OA, but patient adherence to exercise routines is low due to lack of guidance regarding optimal protocols and lack of engagement during the repetitive routines that patients find tedious and boring.

The Knee Biofeedback Rehabilitation Interface for Game-based Home Therapy ("KneeBRIGHT") system combines electromyography (EMG) biofeedback with video game therapy to provide knee OA patients with an engaging, effective tool for conducting rehabilitation exercises at home. KneeBRIGHT aims to motivate patients with knee OA to conduct regular muscle strengthening exercise through an engaging, EMG-driven video game therapy.

Overall goal of the program is to improve knee OA outcomes through effective and motivating rehabilitation exercises. Participants will be randomized to two groups: (1) KneeBRIGHT group; (2) Standard rehabilitation group. Both groups will undergo baseline and follow up assessment to measure the patient-reported outcomes and thigh muscle strength. Participants in both groups will undergo a 12-week program including 3 exercise sessions per week that includes a combination of in-person and at home sessions. Pre and post intervention outcome measures will be compared to explore the effectiveness. Technology acceptance will also be studied in patients randomized to KneeBRIGHT group.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the leading cause of disability in the United States. As osteoarthritis is associated with the lower limb muscle weakness, rehabilitation focused on quadriceps and other lower extremity muscle strengthening is a well-established treatment for patients with knee OA. However, patient adherence to exercise routines is low due to the lack of guidance regarding optimal protocols, and poor engagement during the repetitive routines that patients find tedious and boring.

Long-term goal of this study is to improve knee OA outcomes through effective and motivating rehabilitation exercises. The Knee Biofeedback Rehabilitation Interface for Game-based Home Therapy ("KneeBRIGHT") system combines electromyography (EMG) biofeedback with video game therapy (VGT) to provide knee OA patients with an engaging, effective tool for conducting rehabilitation exercises at home. KneeBRIGHT aims to motivate patients with knee OA to conduct regular muscle strengthening exercise through an engaging, EMG-driven video game therapy.

Participants with age from 40-75, with independent ambulation and with the diagnosis of knee OA made by x-ray and a score of at least 2 (out of 4) on the Kellgren-Lawrence OA radiographic classification system will be included in the study. Participants with psychiatric or cognitive impairment (e.g., dementia), symptomatic spine, hip, ankle, or foot disease other than OA that would interfere with assessment of the knee will be excluded. Participants with balance or vestibular disorders, peripheral neuropathy, skin conditions that prevent EMG electrode placement, prisoner, pregnant women (by report), non-English-speaking, individuals who are visually and/or hearing impaired will also be excluded.

Eligible participants will be randomized to two groups: (1) KneeBRIGHT group; (2) Standard rehabilitation group. Both groups will undergo baseline and follow up assessment to measure the patient-reported outcomes and thigh muscle strength. Participants in both groups will undergo a 12-week program including 3 exercise sessions per week that includes a combination of in-person and at home sessions

Both groups will undergo same rehabilitation protocol which will begin with sessions supervised in the clinic by the study team physical therapist and gradually home sessions will be added. Participants in KneeBRIGHT group will perform the quadriceps strengthening exercises with the video-games based activities. The EMG biofeedback units and video game w/laptop will be provided to the subjects for home use. Subjects will receive instruction on how to apply the EMG biofeedback unit and use of the video game. KneeBRIGHT Game Activities consists of an introduction of the player to the virtual world and the missions, the player customizes the personal avatar and completes a series of calibration contractions and practice exercises to gain familiarity with the game controls. Through the EMG system, a player's muscle contractions translate into physical movements of the avatar and control of vehicles within the virtual environment. Each quest-type challenge is designed to permit play in a seated, supine, supported standing, or freestanding position, based on an individual's physical status. User interactions with the game incorporate knee extension exercises and functional movements that provide optimal therapeutic benefits.

Participants in both groups will undergo combination of home and in clinic sessions. Protocol will start with six clinic visits in order to maximize familiarity with the exercise routines and equipment. Home sessions will be added after 2 weeks in rehabilitation. The sessions will consist of warm up, strengthening, balance, precision and gentle stretching exercises. Strengthening exercises will be focused on quadriceps, hamstring, calf and gluteal muscles. Stretching exercises will be focused on quadriceps, hamstring and calf muscles. Progression will be guided by the rehabilitation principles and participants response to the exercise. The amount of these exercises will depend on how they make the subject feel. The rehabilitation program will allow the subject to increase the amount of exercise they can perform. Exercises will be limited if the subject feels discomfort. Overall, protocol will consist of 36 sessions in total, 20 in clinic sessions and 16 home-based sessions.

Pre and post intervention outcome measures will be compared to explore the effectiveness. Technology acceptance will also be studied in patients randomized to KneeBRIGHT group.

Overall, KneeBRIGHT has the potential to significantly enhance OA rehabilitation by improving functional recovery through physical practice of specific, adaptive exercise and promoting adherence through fun games and performance feedback. Use of the KneeBRIGHT system in teletherapy may increase access to remote/underserved areas and extend the range of existing rehabilitation facilities.

Statistical analysis Knee function assessed by composite KOOS score prior to the study will be compared to the KOOS score recorded post-intervention to test the primary hypothesis that patients conducting the KneeBRIGHT exercise will significantly improve knee function compared to the control group. Pre-intervention KOOS scores measures will be subtracted from the post-intervention scores to produce a set of delta values. These delta values will be analyzed via Analysis of Covariance (ANCOVA). A p≤0.05 decision rule will be utilized as the rejection criterion.

Questionnaire results will be used to test the hypothesis that patients using the KneeBRIGHT system demonstrate increased levels of engagement compared to those conducting a conventional exercise routine. The questionnaire scores will be tallied to produce composite scores. These composite scores will be analyzed via a linear mixed model. A p≤0.05 decision rule will be used as the null hypothesis rejection criterion.

Timing data from the home visits will be analyzed by comparing the minutes of exercise with the KneeBRIGHT system to minutes of exercise with the standard exercise regimen in the control group to test the hypothesis that exercise duration is greater with the KneeBRIGHT system. Mean usage time on each system will be analyzed via Student's paired t-test, with P v≤0.05 as the null hypothesis rejection criterion.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75
* Diagnosis of Osteoarthritis
* Independent ambulation without assistive device

Exclusion Criteria:

* Individuals who have psychiatric or cognitive impairment (e.g., dementia) that interferes with their ability to follow instructions or provide voluntary consent
* Symptomatic spine, hip, ankle, or foot disease other than osteoarthritis that would interfere with assessment of the knee.
* Balance or vestibular disorders
* Peripheral neuropathy
* Skin conditions that prevent EMG electrode placement
* Prisoner
* Pregnant (by report)
* Non-English-speaking
* Individuals who are visually and/or hearing impaired

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Hart, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams RJ, Lichter MD, Krepkovich ET, Ellington A, White M, Diamond PT. Assessing upper extremity motor function in practice of virtual activities of daily living. IEEE Trans Neural Syst Rehabil Eng. 2015 Mar;23(2):287-96. doi: 10.1109/TNSRE.2014.2360149. Epub 2014 Sep 24. PMID 25265612
- [Background] Adams RJ, Lichter MD, Ellington A, White M, Armstead K, Patrie JT, Diamond PT. Virtual Activities of Daily Living for Recovery of Upper Extremity Motor Function. IEEE Trans Neural Syst Rehabil Eng. 2018 Jan;26(1):252-260. doi: 10.1109/TNSRE.2017.2771272. PMID 29324411
- [Background] Adams RJ. Strength and BALance (SABAL) Virtual Trainer. NIA: 1R41AG046958-01A1, 2015.
- [Background] Ardali G. A daily adjustable progressive resistance exercise protocol and functional training to increase quadriceps muscle strength and functional performance in an elderly homebound patient following a total knee arthroplasty. Physiother Theory Pract. 2014 May;30(4):287-97. doi: 10.3109/09593985.2013.868064. Epub 2014 Jan 7. PMID 24397371
- [Background] Babault N, Pousson M, Ballay Y, Van Hoecke J. Activation of human quadriceps femoris during isometric, concentric, and eccentric contractions. J Appl Physiol (1985). 2001 Dec;91(6):2628-34. doi: 10.1152/jappl.2001.91.6.2628. PMID 11717228
- [Background] Bell DR, Guskiewicz KM, Clark MA, Padua DA. Systematic review of the balance error scoring system. Sports Health. 2011 May;3(3):287-95. doi: 10.1177/1941738111403122. PMID 23016020
- [Background] Bennell K, Hinman R. Exercise as a treatment for osteoarthritis. Curr Opin Rheumatol. 2005 Sep;17(5):634-40. doi: 10.1097/01.bor.0000171214.49876.38. PMID 16093845
- [Background] Bitton R. The economic burden of osteoarthritis. Am J Manag Care. 2009 Sep;15(8 Suppl):S230-5. PMID 19817509
- [Background] Bossen D, Buskermolen M, Veenhof C, de Bakker D, Dekker J. Adherence to a web-based physical activity intervention for patients with knee and/or hip osteoarthritis: a mixed method study. J Med Internet Res. 2013 Oct 16;15(10):e223. doi: 10.2196/jmir.2742. PMID 24132044
- [Background] Bossen D, Veenhof C, Van Beek KE, Spreeuwenberg PM, Dekker J, De Bakker DH. Effectiveness of a web-based physical activity intervention in patients with knee and/or hip osteoarthritis: randomized controlled trial. J Med Internet Res. 2013 Nov 22;15(11):e257. doi: 10.2196/jmir.2662. PMID 24269911
- [Background] Cameron C. Patient compliance: recognition of factors involved and suggestions for promoting compliance with therapeutic regimens. J Adv Nurs. 1996 Aug;24(2):244-50. doi: 10.1046/j.1365-2648.1996.01993.x. PMID 8858426
- [Background] Campbell R, Evans M, Tucker M, Quilty B, Dieppe P, Donovan JL. Why don't patients do their exercises? Understanding non-compliance with physiotherapy in patients with osteoarthritis of the knee. J Epidemiol Community Health. 2001 Feb;55(2):132-8. doi: 10.1136/jech.55.2.132. PMID 11154253
- [Background] Carr A. Barriers to the effectiveness of any intervention in OA. Best Pract Res Clin Rheumatol. 2001 Oct;15(4):645-56. doi: 10.1053/berh.2001.0179. PMID 11567545
- [Background] Chen H, Rong W, Ma X, Qu,Y and Xiong Z. An Extended Technology Acceptance Model for MobileSocial Gaming Service Popularity Analysis. Mobile Information Systems, vol. 2017. doi:10.1155/2017/3906953
- [Background] Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S208-28. doi: 10.1002/acr.20632. No abstract available. PMID 22588746
- [Background] Creating healthcare data applications to promote HIPAA and HITECH Compliance. Amazon Web Services. http://aws.amazon.com/compliance/#hipaa
- [Background] Davis FD. Perceived Usefulness, Ease of Use, and User Acceptance of IT. MIS Quarterly. 1989;13(3):319-40.
- [Background] De Luca CJ, Kuznetsov M, Gilmore LD, Roy SH. Inter-electrode spacing of surface EMG sensors: reduction of crosstalk contamination during voluntary contractions. J Biomech. 2012 Feb 2;45(3):555-61. doi: 10.1016/j.jbiomech.2011.11.010. Epub 2011 Dec 9. PMID 22169134
- [Background] Devos-Comby L, Cronan T, Roesch SC. Do exercise and self-management interventions benefit patients with osteoarthritis of the knee? A metaanalytic review. J Rheumatol. 2006 Apr;33(4):744-56. PMID 16583478
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Ericsson YB, Dahlberg LE, Roos EM. Effects of functional exercise training on performance and muscle strength after meniscectomy: a randomized trial. Scand J Med Sci Sports. 2009 Apr;19(2):156-65. doi: 10.1111/j.1600-0838.2008.00794.x. Epub 2008 Apr 6. PMID 18397193
- [Background] Farr JN, Going SB, Lohman TG, Rankin L, Kasle S, Cornett M, Cussler E. Physical activity levels in patients with early knee osteoarthritis measured by accelerometry. Arthritis Rheum. 2008 Sep 15;59(9):1229-36. doi: 10.1002/art.24007. PMID 18759320
- [Background] Farr JN, Going SB, McKnight PE, Kasle S, Cussler EC, Cornett M. Progressive resistance training improves overall physical activity levels in patients with early osteoarthritis of the knee: a randomized controlled trial. Phys Ther. 2010 Mar;90(3):356-66. doi: 10.2522/ptj.20090041. Epub 2010 Jan 7. PMID 20056719
- [Background] Fetscherin M, Lattemann C, User Acceptance of Virtual Worlds. J Electronic Comm Research. 2008; 9(3):231-42.
- [Background] Fisher NM, Gresham G, Pendergast DR. Effects of a quantitative progressive rehabilitation program applied unilaterally to the osteoarthritic knee. Arch Phys Med Rehabil. 1993 Dec;74(12):1319-26. doi: 10.1016/0003-9993(93)90087-q. PMID 8259900
- [Background] Fransen M, McConnell S, Bell M. Therapeutic exercise for people with osteoarthritis of the hip or knee. A systematic review. J Rheumatol. 2002 Aug;29(8):1737-45. PMID 12180738
- [Background] Fransen M, McConnell S. Exercise for osteoarthritis of the knee. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD004376. doi: 10.1002/14651858.CD004376.pub2. PMID 18843657
- [Background] Gell NM, Rosenberg DE, Demiris G, LaCroix AZ, Patel KV. Patterns of technology use among older adults with and without disabilities. Gerontologist. 2015 Jun;55(3):412-21. doi: 10.1093/geront/gnt166. Epub 2013 Dec 30. PMID 24379019
- [Background] Goldman RJ, Reinbold KA, Iglarsh ZA, Neustadter LM, Oatis CA, Schumacher HR. Phase I design and evaluation of an isometric muscle reeducation device for knee osteoarthritis rehabilitation. J Rehabil Res Dev. 2003 Mar-Apr;40(2):95-107. doi: 10.1682/jrrd.2003.03.0095. PMID 15077636
- [Background] Higgins LD, Taylor MK, Park D, Ghodadra N, Marchant M, Pietrobon R, Cook C; International Knee Documentation Committee. Reliability and validity of the International Knee Documentation Committee (IKDC) Subjective Knee Form. Joint Bone Spine. 2007 Dec;74(6):594-9. doi: 10.1016/j.jbspin.2007.01.036. Epub 2007 Aug 6. PMID 17888709
- [Background] Holden RJ, Karsh BT. The technology acceptance model: its past and its future in health care. J Biomed Inform. 2010 Feb;43(1):159-72. doi: 10.1016/j.jbi.2009.07.002. Epub 2009 Jul 15. PMID 19615467
- [Background] Hootman JM, Helmick CG. Projections of US prevalence of arthritis and associated activity limitations. Arthritis Rheum. 2006 Jan;54(1):226-9. doi: 10.1002/art.21562. PMID 16385518
- [Background] Hopkins JT, Ingersoll CD, Krause BA, Edwards JE, Cordova ML. Effect of knee joint effusion on quadriceps and soleus motoneuron pool excitability. Med Sci Sports Exerc. 2001 Jan;33(1):123-6. doi: 10.1097/00005768-200101000-00019. PMID 11194097
- [Background] Hsu JK, Thibodeau R, Wong SJ, Zukiwsky D, Cecile S, Walton DM. A "Wii" bit of fun: the effects of adding Nintendo Wii((R)) Bowling to a standard exercise regimen for residents of long-term care with upper extremity dysfunction. Physiother Theory Pract. 2011 Apr;27(3):185-93. doi: 10.3109/09593985.2010.483267. Epub 2010 Aug 10. PMID 20698793
- [Background] Imoto AM, Peccin MS, Trevisani VF. Quadriceps strengthening exercises are effective in improving pain, function and quality of life in patients with osteoarthritis of the knee. Acta Ortop Bras. 2012;20(3):174-9. doi: 10.1590/S1413-78522012000300008. PMID 24453599
- [Background] Jenkinson CM, Doherty M, Avery AJ, Read A, Taylor MA, Sach TH, Silcocks P, Muir KR. Effects of dietary intervention and quadriceps strengthening exercises on pain and function in overweight people with knee pain: randomised controlled trial. BMJ. 2009 Aug 18;339:b3170. doi: 10.1136/bmj.b3170. PMID 19690345
- [Background] Jones SW, Hill RJ, Krasney PA, O'Conner B, Peirce N, Greenhaff PL. Disuse atrophy and exercise rehabilitation in humans profoundly affects the expression of genes associated with the regulation of skeletal muscle mass. FASEB J. 2004 Jun;18(9):1025-7. doi: 10.1096/fj.03-1228fje. Epub 2004 Apr 14. PMID 15084522
- [Background] Juhl C, Christensen R, Roos EM, Zhang W, Lund H. Impact of exercise type and dose on pain and disability in knee osteoarthritis: a systematic review and meta-regression analysis of randomized controlled trials. Arthritis Rheumatol. 2014 Mar;66(3):622-36. doi: 10.1002/art.38290. PMID 24574223
- [Background] Khaled Takey ,Olfat A. Kandil, and, Shimaa N. Abo Elazm. Isokinetic quadriceps peak torque, average power and total work at different angular knee velocities of physical therapy for internal medicine its surgery and geriatrics , Basic Science Dept. 1, 2,3 Misr University for science and technology.
- [Background] Kijowski R, Blankenbaker D, Stanton P, Fine J, De Smet A. Arthroscopic validation of radiographic grading scales of osteoarthritis of the tibiofemoral joint. AJR Am J Roentgenol. 2006 Sep;187(3):794-9. doi: 10.2214/AJR.05.1123. PMID 16928947
- [Background] Knight KL. Quadriceps strengthening with the DAPRE technique: case studies with neurological implications. Med Sci Sports Exerc. 1985 Dec;17(6):646-50. doi: 10.1249/00005768-198512000-00004. PMID 4079735
- [Background] Lange AK, Vanwanseele B, Fiatarone Singh MA. Strength training for treatment of osteoarthritis of the knee: a systematic review. Arthritis Rheum. 2008 Oct 15;59(10):1488-94. doi: 10.1002/art.24118. PMID 18821647
- [Background] Laferriere P, Lemaire ED, Chan ADC. Surface Electromyographic Signals Using Dry Electrodes. IEEE Trans Ins Meas 60(10): 3259- 3268, 2011.
- [Background] Loeser RF Jr. Aging and the etiopathogenesis and treatment of osteoarthritis. Rheum Dis Clin North Am. 2000 Aug;26(3):547-67. doi: 10.1016/s0889-857x(05)70156-3. PMID 10989512
- [Background] Lucca JA, Recchiuti SJ. Effect of electromyographic biofeedback on an isometric strengthening program. Phys Ther. 1983 Feb;63(2):200-3. doi: 10.1093/ptj/63.2.200. PMID 6823470
- [Background] Lyons GM, Sharma P, Baker M, O'Malley S, Shanahan A, A computer game-based EMG biofeedback system for muscle rehabilitation. Proc 25th Annual International Conference of the IEEE Eng Med Biol Society, 2003, 2:1625 - 8.
- [Background] MarketResearch.com,
- [Background] Marks R. Knee osteoarthritis and exercise adherence: a review. Curr Aging Sci. 2012 Feb;5(1):72-83. doi: 10.2174/1874609811205010072. PMID 21762086
- [Background] McAuley E, Jerome GJ, Elavsky S, Marquez DX, Ramsey SN. Predicting long-term maintenance of physical activity in older adults. Prev Med. 2003 Aug;37(2):110-8. doi: 10.1016/s0091-7435(03)00089-6. PMID 12855210
- [Background] McCreadie C, Tinker A. The acceptability of assistive technology to older people. Ageing and Society 2005;25(1);91-110.
- [Background] Murphy L, Helmick CG. The impact of osteoarthritis in the United States: a population-health perspective: A population-based review of the fourth most common cause of hospitalization in U.S. adults. Orthop Nurs. 2012 Mar-Apr;31(2):85-91. doi: 10.1097/NOR.0b013e31824fcd42. PMID 22446800
- [Background] National Center for Chronic Disease Prevention and Health Promotion. Arthritis: Meeting the Challenge of living well (2013). Report available through: http://www.cdc.gov/chronicdisease/resources/publications/aag/pdf/2013/arthritis-aag-2013_508.pdf
- [Background] Ng GY, Zhang AQ, Li CK. Biofeedback exercise improved the EMG activity ratio of the medial and lateral vasti muscles in subjects with patellofemoral pain syndrome. J Electromyogr Kinesiol. 2008 Feb;18(1):128-33. doi: 10.1016/j.jelekin.2006.08.010. Epub 2006 Oct 27. PMID 17070701
- [Background] Ostir GV, Cohen-Mansfield J, Leveille S, Volpto S and Guralnik JM. The association of positive and negative affect and exercise self-efficacy in older adults. J Aging Phys Act 2003; 11: 265-74.
- [Background] Parker E. A new approach to vision therapy based on naturalistic 3-D computer gaming. NEI: 5R44EY021079-04, 2013.
- [Background] Parker E. A wireless EMG data collection and analysis system. NIAMS: 5R44AR047274-03, 2004.
- [Background] Petersson IF, Boegard T, Saxne T, Silman AJ, Svensson B. Radiographic osteoarthritis of the knee classified by the Ahlback and Kellgren & Lawrence systems for the tibiofemoral joint in people aged 35-54 years with chronic knee pain. Ann Rheum Dis. 1997 Aug;56(8):493-6. doi: 10.1136/ard.56.8.493. PMID 9306873
- [Background] Pisters MF, Veenhof C, Schellevis FG, Twisk JW, Dekker J, De Bakker DH. Exercise adherence improving long-term patient outcome in patients with osteoarthritis of the hip and/or knee. Arthritis Care Res (Hoboken). 2010 Aug;62(8):1087-94. doi: 10.1002/acr.20182. PMID 20235201
- [Background] Piva SR, Fitzgerald GK, Irrgang JJ, Fritz JM, Wisniewski S, McGinty GT, Childs JD, Domenech MA, Jones S, Delitto A. Associates of physical function and pain in patients with patellofemoral pain syndrome. Arch Phys Med Rehabil. 2009 Feb;90(2):285-95. doi: 10.1016/j.apmr.2008.08.214. PMID 19236982
- [Background] Przybylski AK, Weinstein N, Ryan RM, Rigby CS. Having to versus wanting to play: background and consequences of harmonious versus obsessive engagement in video games. Cyberpsychol Behav. 2009 Oct;12(5):485-92. doi: 10.1089/cpb.2009.0083. PMID 19772442
- [Background] Rand D, Kizony R, Weiss PT. The Sony PlayStation II EyeToy: low-cost virtual reality for use in rehabilitation. J Neurol Phys Ther. 2008 Dec;32(4):155-63. doi: 10.1097/NPT.0b013e31818ee779. PMID 19265756
- [Background] Rigby C and Przybylski A. Virtual worlds and the learner hero: How today's video games can inform tomorrow's digital learning environments. Theory and Research in Education. 2009; 7(2):214-23.
- [Background] Rigby, CS, Ryan, RM. Glued to games: How video games draw us in and hold us spellbound. Santa Barbara: Praeger; 2011. 173
- [Background] Risberg MA, Holm I, Tjomsland O, Ljunggren E, Ekeland A. Prospective study of changes in impairments and disabilities after anterior cruciate ligament reconstruction. J Orthop Sports Phys Ther. 1999 Jul;29(7):400-12. doi: 10.2519/jospt.1999.29.7.400. PMID 10416180
- [Background] Ryan, RM, Rigby, CS, Przybylski, AK. Motivation pull of video games: A Self-determination theory approach. Motivation and Emotion 2006; 30:347-365.
- [Background] Schutzer KA, Graves BS. Barriers and motivations to exercise in older adults. Prev Med. 2004 Nov;39(5):1056-61. doi: 10.1016/j.ypmed.2004.04.003. PMID 15475041
- [Background] Hu B, Skou ST, Wise BL, Williams GN, Nevitt MC, Segal NA. Lower Quadriceps Rate of Force Development Is Associated With Worsening Physical Function in Adults With or at Risk for Knee Osteoarthritis: 36-Month Follow-Up Data From the Osteoarthritis Initiative. Arch Phys Med Rehabil. 2018 Jul;99(7):1352-1359. doi: 10.1016/j.apmr.2017.12.027. Epub 2018 Jan 31. PMID 29408538
- [Background] Taylor MJ, McCormick D, Shawis T, Impson R, Griffin M. Activity-promoting gaming systems in exercise and rehabilitation. J Rehabil Res Dev. 2011;48(10):1171-86. doi: 10.1682/jrrd.2010.09.0171. PMID 22234662
- [Background] van Gool CH, Penninx BW, Kempen GI, Rejeski WJ, Miller GD, van Eijk JT, Pahor M, Messier SP. Effects of exercise adherence on physical function among overweight older adults with knee osteoarthritis. Arthritis Rheum. 2005 Feb 15;53(1):24-32. doi: 10.1002/art.20902. PMID 15696558
- [Background] van Linschoten R, van Middelkoop M, Berger MY, Heintjes EM, Verhaar JA, Willemsen SP, Koes BW, Bierma-Zeinstra SM. Supervised exercise therapy versus usual care for patellofemoral pain syndrome: an open label randomised controlled trial. BMJ. 2009 Oct 20;339:b4074. doi: 10.1136/bmj.b4074. PMID 19843565
- [Background] Vincent KR, Vincent HK. Resistance exercise for knee osteoarthritis. PM R. 2012 May;4(5 Suppl):S45-52. doi: 10.1016/j.pmrj.2012.01.019. PMID 22632702
- [Background] Wasielewski NJ, Parker TM, Kotsko KM. Evaluation of electromyographic biofeedback for the quadriceps femoris: a systematic review. J Athl Train. 2011 Sep-Oct;46(5):543-54. doi: 10.4085/1062-6050-46.5.543. PMID 22488142
- [Background] Witvrouw E, Callaghan MJ, Stefanik JJ, Noehren B, Bazett-Jones DM, Willson JD, Earl-Boehm JE, Davis IS, Powers CM, McConnell J, Crossley KM. Patellofemoral pain: consensus statement from the 3rd International Patellofemoral Pain Research Retreat held in Vancouver, September 2013. Br J Sports Med. 2014 Mar;48(6):411-4. doi: 10.1136/bjsports-2014-093450. No abstract available. PMID 24569145
- [Background] Yelin E, Murphy L, Cisternas MG, Foreman AJ, Pasta DJ, Helmick CG. Medical care expenditures and earnings losses among persons with arthritis and other rheumatic conditions in 2003, and comparisons with 1997. Arthritis Rheum. 2007 May;56(5):1397-407. doi: 10.1002/art.22565. PMID 17469096
- [Background] Yilmaz OO, Senocak O, Sahin E, Baydar M, Gulbahar S, Bircan C, Alper S. Efficacy of EMG-biofeedback in knee osteoarthritis. Rheumatol Int. 2010 May;30(7):887-92. doi: 10.1007/s00296-009-1070-9. Epub 2009 Aug 20. PMID 19693508
- See also: Brendon Hall group — http://brandonhall.com/excellence-learning.php?year=2013
- See also: KOOS Questionnaire — http://www.koos.nu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized= 34
Pre-assignment Details: Excluded (n=4) Scheduling reasons=2 The patients refused participation because of pandemic= 2
Groups:
- KneeBright Group: Participants in this group will perform exercises aimed to improve the muscle strength, balance and precision. Participants will perform exercises three times a week for 12 weeks. Each session will last for an hour. Some of the exercises will be performed with the KneeBright Device while playing a video game.
  KneeBright Group: The KneeBRIGHT group will use KneeBright device which consists of an EMG biofeedback interface software that guides users through exercise routines. The wireless EMG sensors includes two small electrodes that will be made to stick to the quadriceps muscles both sides. KneeBRIGHT software features a virtual world wherein patients complete challenges controlling the in-game avatar with the EMG units during exercises specific to knee osteoarthritis rehabilitation.
  The KneeBRIGHT software will incorporates a variety of exercises for strengthening the quadriceps and will employ algorithms based on the Daily Adjustable Progressive Resistance Exercise (DAPRE) technique, in which the quantity of repetitions performed in these sets is then used to determine the appropriate increase (or possibly decrease) in target resistance for the next sets/sessions.
Period: Overall Study
Arm/Group | KneeBright Group | Standard Rehabilitation Group
Started | 17 | 17
Completed | 15 | 14
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Race data were collected at the screening visit. Patients were asked to self-report their individual race identity.
Groups:
- KneeBright Group: Participants in this group will perform exercises aimed to improve the muscle strength, balance and precision. Participants will perform exercises three times a week for 12 weeks. Each session will last for an hour. Some of the exercises will be performed with the KneeBright Device while playing a video game.
  KneeBright Group: The KneeBRIGHT group will use KneeBright device which consists of an EMG biofeedback interface software that guides users through exercise routines. The wireless EMG sensors includes two small electrodes that will be made to stick to the quadriceps muscles both sides. KneeBRIGHT software features a virtual world wherein patients complete challenges controlling the in-game avatar with the EMG units during exercises specific to knee osteoarthritis rehabilitation.
  The KneeBRIGHT software will incorporate a variety of exercises for strengthening the quadriceps and will employ algorithms based on the Daily Adjustable Progressive Resistance Exercise (DAPRE) technique, in which the quantity of repetitions performed in these sets is then used to determine the appropriate increase (or possibly decrease) in target resistance for the next sets/sessions.
- Total: Total of all reporting groups
Arm/Group | KneeBright Group | Standard Rehabilitation Group | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 1 | 10
  >=65 years | 6 | 13 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (4.9) | 63.4 (6.5) | 66.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Subjects were each asked to self-report race identity
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 14 | 14 | 28
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS has 5 subscales: Symptoms, Pain, Sports, Activities of Daily Living (ADL) and quality of life (QOL). Each scale is expressed on a scale from 0-100 points where 100 = best perceived knee function and 0=worst perceived knee function. The outcome of this study is expressed as a change score from pre-post treatment where positive scores indicate an improvement on each KOOS subscale.
Time Frame: KOOS scores will be measured at baseline, day 1 and at the end of intervention, at 12 weeks.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | KneeBright Group | Standard Rehabilitation Group
Number analyzed (Participants) | 15 | 14
score on a scale
  KOOS Symptoms | 3.3 [-.8 to 7.4] | 8.9 [4.7 to 13.2]
  KOOS Pain | 4.6 [-2.2 to 11.5] | 9.7 [2.6 to 16.8]
  KOOS ADL | 6.4 [-.9 to 13.6] | 11.2 [3.7 to 18.8]
  KOOS Sports | 8.7 [-1 to 18.4] | 16.4 [6.4 to 26.5]
  KOOS QOL | 9.2 [1.9 to 16.5] | 9.8 [2.3 to 17.4]
Statistical Analysis 1: Comparison: KneeBright Group vs Standard Rehabilitation Group; The 12-week changes in the KOOS scores, and the 12-week changes in the IKDC scores were analyzed by way of analysis of covariance (ANCOVA). Covariates: Age and sex of the subject, the subject's baseline outcome measure, the subject's baseline IKDC Total score, and the subject's standardized intake date (i.e., i.e., subject's intake date minus the intake date of the first enrolled subject) served as the ANCOVA concomitant adjustment variables; Test type: Superiority; p < 0.05, ANCOVA

2. Secondary Outcome: Change in Peak Torque of Thigh Muscles Strength Testing
Description: Thigh muscle strength will be measured at baseline and follow up. Participants will be asked to perform thigh muscle (quadriceps / knee extension) contractions while measures of strength using a dynamometer (biodex system 4) are recorded. Participants will be asked to perform repeated, maximal muscle contractions to test knee extension muscle strength on the test limb (unilateral test, one thigh tested on each particiant). We recorded peak torque defined as the maximal torque achieved during knee extension contractions. The outcome score is expressed as a change in peak torque from pre-post treatment. Positive numbers indicate increases in strength.
Time Frame: Peak torque (muscle strength) will be measured at baseline, day 1 and at the end of intervention, at 12 weeks.
Population: Data from 4 participants in the KneeBright group and 2 participants from the Standard Rehabilitation group were removed due to bad/unuseable strength data. Therefore, 11 in the kneebright group and 12 in the standard rehab group were included in this analysis.
Measure: Mean (90% Confidence Interval); unit: Nm/kg
Units Other Than Participants: thighs
Arm/Group | KneeBright Group | Standard Rehabilitation Group
Number analyzed (Participants) | 11 | 12
Number analyzed (thighs) | 11 | 12
Nm/kg
  Extension peak torque 90degree | 0.11 [-0.02 to 0.24] | 0.11 [-0.02 to 0.23]
  Extension peak torque 180 degree | 0.07 [-0.13 to 0.27] | -0.06 [-0.25 to 0.13]

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Description: There were no Serious Adverse events recorded during this study
Arm/Group | KneeBright Group | Standard Rehabilitation Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT04187092/Prot_SAP_000.pdf